CLINICAL TRIAL: NCT01000415
Title: Comparing Standard Concurrent Chemo-radiation to Neoadjuvant Chemotherapy Then Surgery or Radiation in Patients Stage Ib2-early IIb Cervical Carcinoma
Brief Title: Comparing Study Between Concurrent Chemoradiation and New Combination Treatment in Cervical Cancer Patients
Acronym: TGOCphaseIII
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thai Gynecologic Oncology Collaborative Group (Network)
Collaborators: National Research Council of Thailand (Other Government); Clinical Research Collaborative Network (Network)
Responsible Party: Thai Gynecologic Oncology Collaborative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGOC-03; ECPSU-522231012
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-03

CONDITIONS: Cervical Cancer
Keywords: Stage Ib2-early IIb of cervical cancer; Neoadjuvant chemotherapy; Cisplatin plus gemcitabine; Radical hysterectomy with pelvic lymphadenectomy; Quality of life; Stage Ib2-IIb of cervical cancer patients
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin plus gemcitabine (Experimental): Experimental arm: neoadjuvant chemotherapy (cisplatin plus gemcitabine) followed by surgery Control arm: concurrent chemoradiation (cisplatin/carboplatin)during standard radiation
  Interventions: Other: Neoadjuvant chemotherapy followed by surgery

INTERVENTIONS:
Other: Neoadjuvant chemotherapy followed by surgery — Cisplatin 50 mg/m2 (in the vein)on day 1 of each 23 day cycle plus gemcitabine 1000 mg/m2 (in the vein) on day 1 and day 8, for 3 cycles: until progression or unacceptable toxicity develops.
  Other Names: Platinol,Platinol-AQ; Gemzar

SUMMARY:
The purpose of this study is:

* to compare the effectiveness between the new strategy of treatment (given cis-platinum plus gemcitabine-neoadjuvant chemotherapy followed by surgery),and standard treatment (given cis-platinum/carboplatin during radiation-concurrent chemoradiation)in specific group of cervical cancer patients (stage Ib2-early IIb)
* to evaluate quality of life in both group of patients(standard treatment vs.experimental group)

DETAILED DESCRIPTION:
According to FIGO classification of cervical cancer, stage Ib2 was classified as clinically visible lesion more than 4.0 cm in greatest dimension and stage IIb was classified tumor invades parametrium must not to pelvic wall. These were the common stages in Thai cervical cancer patients,and made a troublesome effect to Thai women. According to this study,stage early IIb with 1/3 of parametrium involvement. Mostly these two stage was treated with concurrent chemoradiation, challenging the possibility of late sequelae of radiation effect. This specific group of patients can be avoid the referred side effect by using neoadjuvant chemotherapy followed by radical hysterectomy with pelvic lymphadenectomy and para-aortic node sampling in operable cases (at least partial response- PR) and concurrent chemoradiation (CCR) in inoperable cases (less than PR). Due to high risk type of these subspecific group, combination chemotherapy instead of single chemotherapy was used as CCR. However in operable cases with identified poor prognostic factor should be receive post operative radiation as the usual manner.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer patients with FIGO stage Ib2-early IIb
* Pathological proven squamous cell carcinoma or adenocarcinoma or adenosquamous cell carcinoma
* ECOG performance status 0-1
* No previous treatment for cervical cancer
* Acceptable hematological,renal,liver function

Exclusion Criteria:

* Previous history of cancer
* Underlying disease not fit for surgery
* Psychological problem
* Obvious pelvic/para-aortic node involvement
* Pregnancy
* HIV positive
* History of bowel obstruction

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 824 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-09 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival comparison between experimental treatment group and standard treatment group | 9 Years

SECONDARY OUTCOMES:
Comparing disease free survival between experimental treatment group and standard treatment group | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Saibua B. Chichareon, MD., Principal Investigator — Thai Gynecologic Oncology Collaborative Group (TGOC)
Locations (1):
- Gynecologic Oncology Unit, Department of Obstertrics and Gynecology, Faculty of medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Termrungruanglert W, Tresukosol D, Vasuratna A, Sittisomwong T, Lertkhachonsuk R, Sirisabya N. Neoadjuvant gemcitabine and cisplatin followed by radical surgery in (bulky) squamous cell carcinoma of cervix stage IB2. Gynecol Oncol. 2005 May;97(2):576-81. doi: 10.1016/j.ygyno.2005.01.048. PMID 15863162